CLINICAL TRIAL: NCT00930189
Title: Randomized, Double Blind, Controlled Study With Verteporfin Photodynamic Therapy And Intravitreal Triamcinolone(IVTA) Vs Triple Therapy With Verteporfin Photodynamic Therapy, Intravitreal Triamcinolone And Intravitreal Ranibizumab In Patients With Subfoveal Choroidal Neovascularization(CNV) Secondary To Age-related Macular Degeneration(AMD)
Brief Title: Comparative Study With Photodynamic Therapy And Triamcinolone Versus Photodynamic Therapy, Triamcinolone And Ranibizumab In Patients With Subfoveal Choroidal Neovascularization
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: Centro Medico Issemym (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APEC-0031
Record Dates: First submitted 2006-12-01; First posted 2009-06-30 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Subfoveal Choroidal Neovascularization
Keywords: age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Photochemotherapy

INTERVENTIONS:
Drug: intravitreal injection of ranibizumab
Drug: intravitreal injection of triamcinolone
Procedure: photodynamic therapy

SUMMARY:
The purpose of this study is to compare the efficacy of photodynamic therapy with verteporfin (PDT) and IVTA vs triple therapy (TT) in patients with subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

The investigators designed a prospective, comparative, randomized, double blind, controlled study. 15 patients with classic subfoveal choroidal neovascularization secondary to age-related macular degeneration were randomized. Triple therapy can potentially offer a new treatment modality for choroidal neovascularization in patients with macular degeneration and other diseases.

DETAILED DESCRIPTION:
Purpose: To compare the efficacy of photodynamic therapy with verteporfin (PDT) and IVTA vs triple therapy (TT) in patients with subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

Methods: Prospective, comparative, randomized, double blind, controlled study. 15 patients with classic subfoveal choroidal neovascularization secondary to age-related macular degeneration were randomized. Group 1: receive PDT followed by 4 mg IVTA (n=7) or group 2: TT (triple Therapy) PDT followed by 4 mg IVTA + 0.5 mg Ranibizumab (n=8).The main outcome measures were visual acuity (VA), mean change in lesion size, mean change in foveal thickness, retreatment rate and the incidence and severity of adverse events.

Results: At 6 months 5 of 7 patients (71.4%) of group 1 and 8 of 8 patients (100% ) of group 2 had lost fewer than 15 letters (P<.001). Three patients (37.5%) of group 2 had an improvement of 3 lines or more. Lesion type, patient age, and lesion size had no influence on the outcome, but baseline VA had a statistically significant effect (P =.006). The median number of treatments in both groups was one. The 28% of PDT-triamcinolone group and 25% of triple therapy group had an increase in intraocular pressure (IOP) that required therapy. Progression or development of cataract was observed in 14.2 % in PDT- IVTA group and 12.5% in Triple therapy group. There were no cases of endophthalmitis. No cardiac or cerebrovascular accidents where presented.

Conclusions: The combination of PDT, intravitreal triamcinolone acetonide and intravitreal ranibizumab is a safe treatment option for neovascular AMD and prevents a considerable decrease in VA. In our patients it seems to be superior than combinated therapy with PDT and triamcinolone.

Clinical Relevance: Triple therapy can potentially offer a new treatment modality for choroidal neovascularization in patients with macular degeneration and other diseases.

:

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD)
* Any visual acuity

Exclusion Criteria:

* Previous treatment
* Glaucoma

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The main outcome measures were visual acuity (VA)
mean change in lesion size
mean change in foveal thickness

SECONDARY OUTCOMES:
retreatment rate
the incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Romero, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Centro Medico Isemmym, Metepec, State of Mexico, Mexico

REFERENCES:
- [Background] Arias L, Garcia-Arumi J, Ramon JM, Badia M, Rubio M, Pujol O. Photodynamic therapy with intravitreal triamcinolone in predominantly classic choroidal neovascularization: one-year results of a randomized study. Ophthalmology. 2006 Dec;113(12):2243-50. doi: 10.1016/j.ophtha.2006.04.039. Epub 2006 Sep 25. PMID 16996600